CLINICAL TRIAL: NCT06645886
Title: A Phase 1/1b, Open-label, Multicenter, Dose Escalation and Dose Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of KQB198 as Monotherapy and in Combination With Anticancer Agents in Participants With Advanced Hematologic Malignancies
Brief Title: A Study to Investigate the Safety and Efficacy of KQB198 as Monotherapy and in Combination in Participants With Advanced Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kumquat Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQB198-102
Record Dates: First submitted 2024-10-02; First posted 2024-10-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancies; Adult
Keywords: CML; dasatinib
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: KQB198
- Combo Therapy Dose Escalation (Experimental)
  Interventions: Drug: KQB198; Drug: Dasatinib
- Combo Therapy Dose Expansion - RP2D (Experimental)
  Interventions: Drug: KQB198; Drug: Dasatinib
- Combo Therapy Dose Expansion - RP2D-1 (Experimental)
  Interventions: Drug: KQB198; Drug: Dasatinib
- Monotherapy Dose Expansion - RP2D (Experimental)
  Interventions: Drug: KQB198
- Monotherapy Dose Expansion - RP2D -1 (Experimental)
  Interventions: Drug: KQB198

INTERVENTIONS:
Drug: KQB198 — Oral KQB198
Drug: Dasatinib — Oral dasatinib
  Arms: Combo Therapy Dose Escalation; Combo Therapy Dose Expansion - RP2D; Combo Therapy Dose Expansion - RP2D-1

SUMMARY:
The goal of this clinical trial is to learn if KQB198 works to treat advanced hematologic malignancies in adults. It will also learn about the safety of KQB198. The main questions it aims to answer are:

* What is the safe dose of KQB198 by itself or in combination with other anti-cancer drugs?
* Does KQB198 alone or in combination with other anti-cancer drugs decrease the size of the tumor?
* What happens to KQB198 in the body?

Participants will:

* Take KQB198 daily, alone or in combination with another anti-cancer drug
* Visit the clinic about 8 times in the first 8 weeks, and then once every 4 weeks after that

ELIGIBILITY:
Inclusion Criteria:

* Adequate organ function

Part 1 and Part 2, Cohort B Participants Only:

• Ph+ CML in chronic phase who have been previously treated with at least 2 different tyrosine kinase inhibitors (TKIs) and are relapsed from or intolerant to those TKIs and ineligible for alternative therapeutic options likely to produce clinical benefit as determined by the investigator.

Part 2, Cohort A Participants Only:

• Participants with Ph+ CML in chronic phase who are on dasatinib prior to study entry and have a warning or failure to dasatinib as determined by the investigator per ELN 2020 guidelines

Exclusion Criteria:

* CML in accelerated or blast phase
* Prior therapy with a similar mechanism of action to KQB198
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of study treatment or result in inability to swallow
* History of interstitial lung disease
* Cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience treatment-emergent adverse events, serious adverse events, and dose-limiting toxicities (Part 1) | 28 Days
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of AEs, SAEs, and DLTs, from first dose of study treatment to 28 days after last dose of study treatment.
Recommended Phase 2 Dose (RP2D) (Part 1) | Up to 30 months
  Evaluate safety and assess number of patients with dose-limiting toxicity to determine the RP2D.
Efficacy of study treatment and optimal biologic dose, as measured by molecular response (MR) per European Leukemia Network (ELN) 2020 Guidelines (Part 2). | Up to 6 Months
  Molecular response is the percentage of BCR-ABL fusion protein found in blood. Calculation of molecular response in Part 2 Cohort A will be the proportion of subjects that experience molecular response 4 (MR4) during the time period from 1st dose of study treatment until 6 months of study treatment. Calculation of molecular response in part 2 cohort B will be the proportion of subjects that experience molecular response 3 (MR3) during the time period from 1st dose of study treatment until 6 months of study treatment.

SECONDARY OUTCOMES:
Efficacy of Study Treatment | Up to 30 months
  Efficacy of study treatment as measured by molecular response (MR) at 3, 6, 9, and 12 months, and anytime.
Efficacy of Study Treatment | Up to 30 Months
  Efficacy of study treatment as measured by duration of response (DOR). DOR is defined as the time from the date when the response is first observed till the date the response is lost or death, whichever is earlier.
Efficacy of Study Treatment | Up to 30 months
  Efficacy of study treatment as measured by time to response (TTR). Response assessments will be summarized by all reported response categories at each visit.
Number of patients who experience treatment-emergent adverse events, serious adverse events, and dose-limiting toxicities (Part 2) | 28 Days After Last Dose
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of AEs, SAEs from first dose of study treatment to 28 days after last dose of study treatment.
Concentration-Time Curve (AUC) | Up to 30 months
Maximum Plasma Concentration (Cmax) | Up to 30 months
Time to Maximum Plasma Concentration (tmax) | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (29):
- United States (10):
  - University of California, San Francisco (UCSF), San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Oncology Hematology Cincinnati, Cincinnati, Ohio
  - Sarah Cannon Research Institute (SCRI) - Transplant and Cellular Therapy Operations, Nashville, Tennessee
  - Texas Oncology Austin Central, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- France (2):
  - CHRU de Tours - Hopital Bretonneau, Tours, Centre-Val de Loire
  - AP-HM - Hopital de la Timone, Marseille
- Germany (2):
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Universitaetsklinikum Jena, Jena, Thuringia
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant Orsola, Bologna, Bologna
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome, Lazio
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Milan, Lombardy
- Stichting Radboud Universitair Medisch Centrum, Nijmegen, Gelderland, Netherlands
- Poland (4):
  - Aidport Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Copernicus PL Sp. z o.o., Wojewodzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
- Spain (4):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Institut Catala d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
- United Kingdom (2):
  - Hammersmith Hospital, London, Greater London
  - Nottingham University Hospitals, Nottingham, Nottinghamshire